CLINICAL TRIAL: NCT01197768
Title: A Multi-Component Behavioral Nutrition Intervention for Homebound Older Adults
Brief Title: A Multi-Component Behavioral Nutrition Intervention for Homebound Elderly
Acronym: MCBNIHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Duke University (Other); Mayo Clinic (Other)
Responsible Party: Principal Investigator, Julie Locher, PhD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F080428013
Record Dates: First submitted 2010-09-02; First posted 2010-09-09 (Estimated); Last update posted 2011-10-14 (Estimated); Status verified 2011-10

CONDITIONS: Undernutrition
MeSH Terms: conditions — Malnutrition | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Nutrition Intervention (Experimental): The intervention group will receive a full nutrition assessment and a nutrition intervention.
  Interventions: Behavioral: Nutrition Intervention
- Control (No Intervention): This group will receive the nutrition assessment but no intervention from a Registered Dietician. If participant appears to be in danger due to BMI or Caloric intake status, their primary care physician will be notified.

INTERVENTIONS:
Behavioral: Nutrition Intervention — Participants randomized to the intervention group receive a comprehensive nutrition assessment and a in-home intervention with follow-up calls from a Registered Dietician who will addresses their risk for becoming under-nourished at multiple levels.
  Arms: Nutrition Intervention

SUMMARY:
The purpose of this study is to evaluate the efficacy and feasibility of a multi-level self-management intervention to improve nutritional intake in a group of homebound older adults (HOAs) who are at especially high risk for undernutrition. The study will be guided by the theoretical approaches of the Ecological Model and Social Cognitive Theory and will use a prospective randomized controlled design to estimate whether individually tailored counseling focusing on social and behavioral aspects of eating results in increased caloric intake and improved nutrition-related health outcomes in a sample of 104 HOAs. The investigators hypothesize that intervention at these levels will improve caloric intake and indirectly improve health outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. at least 65 years of age
2. homebound (based upon Medicare's definition of homebound status)
3. able to communicate or have a caregiver who is able to communicate
4. living in a private residence
5. experiencing either an acute illness or chronic condition
6. not consuming enough calories to maintain body weight or weight loss of > 5% over past 6 months (if known)

Exclusion Criteria:

1. significantly cognitive impaired (MMSE < 24 if living alone or MMSE < 15 if living with caregiver) (if known)
2. terminally ill
3. any cancer diagnosis within the past five years (melanoma excluded)
4. end-stage renal disease
5. gastric or enteral tube-feedings
6. dependent on a ventilator

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2008-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Caloric Intake | 2 and 8 months post-baseline
  At each of the data collection points, (3) 24 hour Food Recalls will be collected and measured against each other. Participants who receive the intervention are hypothesized to increase their caloric intake post-baseline.

SECONDARY OUTCOMES:
Health services utilization, specifically hospitalization and re-hospitalization | 6 months from follow-up assessment
  Patients receiving the intervention are hypothesized to have lower rates of hospitalization and re-hospitalization due to increased caloric intake and a reduced rate of physical decline.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States